CLINICAL TRIAL: NCT05266274
Title: A Single-center, Single-arm Clinical Study of the Clinical Efficacy and Safety of CD47 Monoclonal Antibody Combined With Azacitidine in the Treatment of Recurrent AML After Transplantation
Brief Title: Clinical Efficacy and Safety of CD47 Monoclonal Antibody Combined With Azacitidine in the Treatment of Recurrent AML After Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI188Y103
Record Dates: First submitted 2022-01-17; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-12

CONDITIONS: Patients With Recurrent Acute Myelogenous Leukemia After Transplantation
MeSH Terms: interventions — Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Treatment of Recurrent AML After Transplantation (Experimental)
  Interventions: Drug: CD47 monoclonal antibody

INTERVENTIONS:
Drug: CD47 monoclonal antibody — patients who meet the criteria are selected, CD47 monoclonal antibody combined with azacitidine is used for the treatment of patients with recurrent AML after transplantation
  Other Names: azacitidine

SUMMARY:
After screening according to the criteria for selection and exclusion, patients who meet the criteria are selected, CD47 monoclonal antibody combined with azacitidine is used for the treatment of patients with recurrent AML after transplantation. The primary outcome is objective response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years old
2. Diagnosis of AML and MDS recurrence after allogeneic hematopoietic stem cell transplantation according to WHO diagnostic criteria (flow MRD≥1%)
3. ECOG rating 0-3
4. Leukocyte ≤ 20×10^9/L (allowing hydroxyurea to lower leukocyte therapy); HB ≥ 70g/L, platelet ≥ 30×10^9/L (allow blood transfusion or supportive therapy such as erythropoietin/thrombopoietin, for those who have met all inclusion criteria but hemoglobin and/or platelet count are not fulfilled, discussion with the sponsor is required to determine the eligibility of the subject based on his/her risk and benefit)
5. Liver function: total bilirubin ≦ 1.5 x ULN; alanine aminotransferase ≦ 3 x ULN; aspartate aminotransferase ≦ 3 x ULN; (except for leukemia infiltration)
6. Renal function: endogenous creatinine clearance ≧60ml/min
7. the international normalized ratio ≤ 1.5, and the prothrombin time or activated partial thromboplastin time ≤ 1.5 × ULN
8. Tolerate bone marrow puncture and undergo the test at the time point required by the program
9. Patients who sign the informed consent form must have the ability to understand and be willing to participate in this study, and sign the informed consent form at the same time.

Exclusion Criteria:

1. Active aGVHD.
2. Patients with a history of myeloproliferative disorders (including myelofibrosis, essential thrombocythemia, polycythemia vera, chronic myeloid leukemia) or with BCR-ABL1 translocation
3. Concomitant central nervous system leukemia
4. Previous history of chronic hemolytic anemia or Coomb test (+) during the screening period
5. Patients who were allergic to azacytidine or CD47 inhibitors or experienced serious adverse reactions because of azacytidine or CD47 inhibitors
6. Simultaneous participation in another interventional clinical study, except for: only participate in an observational (non-interventional) clinical study; in the survival follow-up phase of an interventional study
7. Glucocorticoids for therapeutic purposes have been used within 7 days prior to the first treatment. Nasal spraying, inhalational, topical glucocorticoids or low-dose intravenous glucocorticoids (i.e., no more than 10 mg/day prednisone or equivalent doses) are permitted. Prophylactic use of glucocorticoids is permitted to avoid allergic reactions from medical interventions (e.g., intravenous contrast gents, chemotherapeutic drugs, or blood transfusions)
8. Live attenuated vaccines within 4 weeks prior to the first day of the study or planned for the treatment period, have undergone major surgical procedures (craniotomy, thoracic or open surgery) or are expected to receive major surgeries during the treatment period (except for PICC and deep vein catheterization)
9. Patients who have non-hematologic toxicity caused by previous anti-leukemia treatment and the toxicity is not returned to NCI CTCAE v5.0 grade 0 to 1 (except for hair loss, fatigue), have uncontrolled active bleeding, coagulation disorders, or require therapeutic treatment with anticoagulants (such as warfarin, low molecular weight heparin, antiplatelet drugs, etc.)
10. Presence of an active or suspected autoimmune disease or a history of the disease in recent 2 years (except for vitiligo, psoriasis, Hashimoto's thyroiditis or Grave's disease that do not require a systemic treatment within the last 2 years, hypothyroidism that only requires thyroid hormone replacement therapy, or type 1 diabetic subjects requiring only insulin therapy)
11. A history of primary immunodeficiency
12. A history of primary immunodeficiency
13. Uncontrolled concurrent diseases include, but are not limited to:

    HIV infection (HIV antibody positive); Severe infections; Symptomatic congestive heart failure (New York Heart Association Grade II to IV) or poorly controlled arrhythmias that may pose a serious risk of cardiac arrest; Arterial hypertension (systolic blood pressure ≥ 160 mmHg or diastolic ≥ 100 mmHg) even with standardized treatment; Any arterial thromboembolic events, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, occurred within 6 months prior to enrollment; History of deep vein thrombosis, pulmonary embolism, or any other severe thromboembolism within 6 months prior to enrollment; Any life-threatening bleeding events such as intracranial hemorrhage or grade 3 or 4 gastrointestinal/variceal bleeding events requiring transfusion, endoscopic or surgical treatment occurred within 6 months prior to enrollment; Subjects with evidence of portal hypertension or previous history of varicose vein bleeding; A history of gastrointestinal perforation and/or fistula within 6 months prior to enrollment.

    Uncontrolled metabolic disorders or other non-malignant systemic diseases that lead to a higher risk and/or uncertainty in survival evaluation.

    Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh grade B or more severe liver cirrhosis.

    History of intestinal obstruction or the following: inflammatory bowel disease or extensive bowel resection, Crohn's disease, ulcerative colitis, or chronic diarrhea.

    Other acute or chronic illnesses, psychiatric disorders, or abnormal laboratory test values that may result in poor adherence or increased risk associated with drug administration, or interference with the interpretation of study results, and who, based on investigator's judgment, are classified as ineligible for this study.

    Acute or chronic active hepatitis B or C infection: HbsAg and/or HbcAb positive and HBV DNA above the upper limit of normal, HBV DNA is not within the normal range after treatment, hepatitis C virus (HCV) antibody positive and RNA positive
14. Patients with any kind of post-transplant complications: veno-occlusive disease (VOD), idiopathic pneumonia syndrome (IPS), septic shock, thrombotic microangiopathy (TMA)
15. A history of other primary malignant tumors
16. Patients with heart failure grade 2 or above
17. Expected survival < 3 months
18. Pregnant or lactating patients
19. Refusal to enroll in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate | about 3 months
  Including complete response/complete response rate of incomplete hematologic recovery /partial response rate（CR/CRi/PR），after each course of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology, Suzhou, Jiangsu, China